CLINICAL TRIAL: NCT05372692
Title: Early-stage Clinical Study of Mesothelin-specific Chimericantigen Receptor T Cells (LD013) in Subjects With Refractory or Relapsed Mesothelin -Positive Ovarian Cancer
Brief Title: Study of LD013 in Subjects With Refractory or Relapsed Mesothelin -Positive Ovarian Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weijia Fang, MD (Other)
Collaborators: Nanjing Blue Shield Biotech Co.,Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Weijia Fang, MD, chief physician, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZhaoPeng
Record Dates: First submitted 2022-05-09; First posted 2022-05-13 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm open clinical study (Experimental): After blood collection from qualified subjects, lymphocytes will be pretreated，the subjects will then be treated with CAR T cells.
  Interventions: Drug: mesothelin-specific chimeric antigen receptor T cell injection

INTERVENTIONS:
Drug: mesothelin-specific chimeric antigen receptor T cell injection — Autologous T cell injection
  Other Names: LD013

SUMMARY:
Early-stage Clinical Study of mesothelin-specific Chimericantigen Receptor T Cells (LD013) in Subjects With Refractory or Relapsed mesothelin-positive Ovarian Cancer

DETAILED DESCRIPTION:
This is a single-arm, open, dose-increasing, and extended early-stage clinical study of mesothin-specific chimeric antigen receptor T cells (LD013) in patients with mesothelin-positive drug-resistant relapsed ovarian cancer. This study included two phases: dose escalation and extension.

ELIGIBILITY:
Inclusion Criteria:

Fully understand and voluntarily sign informed consent.

* Aged at least 18 years old，female.
* Expected survival > 12weeks.
* Eastern Cooperative Oncology Group (ECOG) score 0or1.
* Staining of mesothelin must be greater than 50% of the cells in the tumor tissue and with apparent expression in the membrane. Tissue obtained for the biopsy must be ≤2year prior to enrollment for screening, not have been previously irradiated or exposed to chemotherapy. If unavailable, new tissue material from a recently obtained surgical or diagnostic biopsy is mandatory for this trial；

Exclusion Criteria:

* Prior treatment with any CART therapy targeting any target.
* Subjects with severe mental disorders.
* Subjects with other malignant tumors.
* Patient is positive for Syphilis, Human Immunodeficiency Virus (HIV) , active Hepatitis B (HBsAg reactive) or Hepatitis C (HCV RNA (qualitative) is detected).
* Detectable clinically relevant central nervous system (CNS) metastases and/or pathology such as epilepsy/seizure, brain Ischemia/ hemorrhage, dementia, cerebellar disease, or autoimmune disease affecting central nervous system；
* Patients with ongoing or active infection.
* Subjects not appropriate to participate in this clinical study judged by investigators.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Early-stage Clinical Study of mesothelin-specific Chimericantigen Receptor T Cells (LD013) in Subjects With Refractory or Relapsed mesothelin-positive Ovarian Cancer
Enrollment: 3 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
objective remission rate | 4-6weeks
  objective remission rate

CONTACTS AND LOCATIONS:
Locations (1):
- First affiliated hospital, School of Medicine, Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen J, Zhao L, Li W, Wang S, Li J, Lv Z, Zhao Y, Liang J, Hu Z, Pan F, He L, Gu L, Guo Z. Glutamine-driven metabolic reprogramming promotes CAR-T cell function through mTOR-SREBP2 mediated HMGCS1 upregulation in ovarian cancer. J Transl Med. 2025 Jul 17;23(1):803. doi: 10.1186/s12967-025-06853-0. PMID 40676647